CLINICAL TRIAL: NCT01121783
Title: Study of the Effect of Lactisole on the Responses to Intragastric Glucose Solution
Brief Title: The Effect of Lactisole on the Responses to Glucose Solution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Northern Care Alliance NHS Foundation Trust (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Mohammed Zubair, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Lactisole
Record Dates: First submitted 2010-05-10; First posted 2010-05-12 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2010-03

CONDITIONS: Blood Glucose; Appetite; Therapeutic Uses; Hormones
MeSH Terms: interventions — lactisole

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- Lactisole-Glucose (Active Comparator)
  Interventions: Other: Lactisole
- Lactisole-water (Active Comparator)
  Interventions: Dietary Supplement: Lactisole
- Water-Glcuose (Placebo Comparator)
  Interventions: Dietary Supplement: Lactisole
- Water-Water (Placebo Comparator)
  Interventions: Dietary Supplement: Lactisole

INTERVENTIONS:
Other: Lactisole — A pre-infusion of lactisole solution (0.25mg/ml) is administered as a bolus (1ml/kg bodyweight)via intragastric tube. After 15 minutes a 1M glucose solution is administered as a bolus via intragastric tube.
  Arms: Lactisole-Glucose
Dietary Supplement: Lactisole — A pre-infusion of lactisole solution (0.25mg/ml)is administered as a bolus (1ml/kg body weight) via intragastric tube. After 15 minutes tap water will be administered as a bolus via the intragastric tube.
  Arms: Lactisole-water
Dietary Supplement: Lactisole — A pre-infusion of tap water(is administered as a bolus (1ml/kg bodyweight)via intragastric tube. After 15 minutes a 1M glucose solution is administered as a bolus via intragastric tube.
  Arms: Water-Glcuose
Dietary Supplement: Lactisole — A pre-infusion of tap water is administered as a bolus (1ml/kg bodyweight)via intragastric tube. After 15 minutes tap water is administered as a bolus via intragastric tube.
  Arms: Water-Water

SUMMARY:
The purpose of the study is to determine whether the sweet taste receptors in the gut are involved in sensing sweet substances and controlling appetite and the amount we eat. Lactisole is a substance commonly used in food products to reduce the perceived sweetness of certain sugars and sweeteners. The aim of this study is to investigate whether the responses to a glucose solution, intragastrically administered to healthy male and female volunteers, is affected by the presence of lactisole in the gut. Understanding the mechanisms by which nutrients are initially detected in the gut and how they influence food intake is critical to the development of novel food products that could reduce food consumption.

DETAILED DESCRIPTION:
Obesity is epidemically prevalent and a major risk factor for chronic diseases making it fundamental to understand the pathways controlling food intake. During the course of a meal and afterwards the gut and brain communicate to control how full the eater feels and thus control the amount of food eaten. The information relayed from the gut to the brain regarding ingested nutrients is of increasing importance and understanding the mechanisms by which nutrient molecules are initially detected in the gut and how they signal to the brain to influence food intake is critical to the development of novel food products that could induce fullness and reduce food consumption. Increasing our understanding of how nutrients are sensed in the gut and how this may influence subsequent food intake provides promising targets for obesity prevention and treatment. Recent discoveries have shown that sweet taste receptors similar to those located in the tongue are present in the gut. It is suggested that theses receptors are involved in the way nutrients are sensed and may play an important role in appetite control and food intake.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18-45 years
* BMI between 18-25kg/m2
* General good health

Exclusion Criteria:

* Underweight or Overweight (Body Mass Index <19 or >25 kg.m-2)
* Females who are pregnant or breastfeeding
* Currently taking medication (except females taking oral contraceptive)
* Smokers
* Currently dieting or have experienced a weight change +/- 3kg in past 6 months
* Metabolic disorders (eg. Type 2 diabetes)
* History of gastrointestinal disorders
* Participation in other research in past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Blood glucose | Blood samples will be collected at baseline and 5, 15 and 30 minute intervals until 150 minutes after the glucose infusion

SECONDARY OUTCOMES:
Subjective appetite ratings | 30 minute intervals
  Participants will be asked to complete visual analogue scale questionnaire (VAS) up to a total of 6 times for the duration of each study
Gastric emptying rate | Breath samples are collected at 5, 15 and 30 minute intervals up to a total of 10 times until 150 minutes
  In order to assess gastric emptying, a stable isotope of carbon, in the form of 13Csodium acetate will be added to the test meal. This is absorbed only once it has passed through the stomach into the duodenum. It is then metabolised and exhaled in the breath as 13Clabelled carbon dioxide (CO2) where it can be measured.
Energy intake
  Energy intake will be assessed by an ad libitum test meal provided at the end of each study and food diaries completed for the remainder of the day
Gut hormones | Blood samples will be collected at baseline, 5, 15 and 30 minute intervals until 150 minutes after glucose infusion.
  Blood samples will be processed to examine hormone levels of GLP-1, PYY, and insulin.

CONTACTS AND LOCATIONS:
Overall Officials: David Thompson, FRCP, fMedSci,, Principal Investigator — University of Manchester
Locations (1):
- Salford Royal NHS Foundation Trust, Manchester, United Kingdom